CLINICAL TRIAL: NCT03810690
Title: A Global, Phase 1/2, Open Label, Dose Escalation Study to Evaluate the Safety, Pharmacodynamics, and Pharmacokinetics of mRNA-3704 in Patients With Isolated Methylmalonic Acidemia Due to Methylmalonyl-CoA Mutase Deficiency
Brief Title: Open Label Study of mRNA-3704 in Patients With Isolated Methylmalonic Acidemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated before the start of dosing due to a business decision and not due to safety or efficacy reasons.
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: mRNA-3704-P101
Record Dates: First submitted 2019-01-14; First posted 2019-01-22 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Methylmalonic Acidemia (MMA); Metabolism, Inborn Errors
MeSH Terms: conditions — Methylmalonic acidemia; Metabolism, Inborn Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation Phase: Dose Level 1 (Experimental): mRNA-3704
  Interventions: Biological: mRNA-3704
- Dose Escalation Phase: Dose Level 2 (Experimental): mRNA-3704
  Interventions: Biological: mRNA-3704
- Dose Escalation Phase: Dose Level 3 (Experimental): mRNA-3704
  Interventions: Biological: mRNA-3704
- Dose Escalation Phase: Dose Level 4 (optional) (Experimental): mRNA-3704
  Interventions: Biological: mRNA-3704
- Dose Expansion Phase: mRNA-3704 (Experimental)
  Interventions: Biological: mRNA-3704

INTERVENTIONS:
Biological: mRNA-3704 — mRNA-3704 dispersion for intravenous (IV) infusion

SUMMARY:
This First-in-Human (FIH) Phase 1/2 study will evaluate mRNA-3704 in patients with methylmalonic acidemia/aciduria (MMA) due to methylmalonyl-coenzyme A mutase (MUT) deficiency between 1 to 18 years of age with elevated plasma methylmalonic acid. The study is designed to characterize baseline biomarker levels followed by assessment of safety, pharmacokinetics, and pharmacodynamics of different doses of mRNA-3704 in patients affected by MMA as part of the Dose Escalation phase.

During the Dose Escalation phase, three dose levels of mRNA-3704 are planned to be investigated in this study among patients with MMA due to MUT deficiency: low dose, mid dose, and high dose. An additional cohort to evaluate a fourth dose level may be considered jointly by the independent SMC and the Sponsor.

Upon establishment of a dose with acceptable safety and pharmacodynamic activity, additional patients will be enrolled in a Dose Expansion phase to allow for further characterization of the safety and pharmacodynamics of mRNA-3704.

Patients in both phases of study will participate in a pre-dosing observational period, followed by a treatment period, and then a follow-up period after withdrawal of treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if all of the following criteria apply:

* Confirmed diagnosis of isolated MMA due to MUT deficiency based on the following criteria:

  * Elevated plasma methylmalonic acid concentrations (≥ 100 µmol/L)
  * Presence of normal serum/plasma Vitamin B12 and plasma homocysteine levels
  * Confirmed diagnosis by molecular genetic testing
* Patient must be ≥ 1 year of age at the time of consent/assent (Inclusion of the first three patients will be restricted to individuals age ≥ 8 years)

Exclusion Criteria:

Patients are excluded from the study if any of the following criteria apply:

* Diagnosis of isolated MMA cblA, cblB, or cblD enzymatic subtypes or methylmalonyl-CoA epimerase deficiency or combined MMA with homocystinuria
* History of organ transplantation
* Previously received gene therapy for the treatment of MMA.
* Estimated glomerular filtration rate (GFR) < 30 mL/min/1.73 m2; or patients who receive chronic dialysis

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Day 1 (initial mRNA-3704 dose) through 52 weeks after final mRNA-3704 dose
Change in plasma methylmalonic acid levels | Week -4 through 36 weeks after initial mRNA-3704 dose
  Baseline (pre-dose levels) to post-dose levels measured after single and after repeated administrations of mRNA-3704

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) after administration of mRNA-3704 | Baseline through 36 weeks after initial mRNA-3704 dose
Time of Cmax (Tmax) | Baseline through 36 weeks after initial mRNA-3704 dose
Area under the plasma concentration-time curve (AUC) | Baseline through 36 weeks after initial mRNA-3704 dose
Change in plasma 2-methylcitrate levels | Week -4 through 36 weeks after initial mRNA-3704 dose
  Baseline (pre-dose levels) to levels measured after single and after repeated administrations of mRNA-3704
Measurement of anti-PEG antibodies | Pre-dose through up to 52 weeks after final mRNA-3704 dose

IPD SHARING:
Plan to Share IPD: No